CLINICAL TRIAL: NCT04334564
Title: Effect of Ginkgo Biloba Capsule on Visual Function of Primary Open-angle Glaucoma With Blood Stasis Syndrome: a Randomized, Double-blind, Placebo Parallel Control, Multicenter Clinical Trial
Brief Title: Effect of Ginkgo Biloba Capsule on Visual Function of Primary Open-angle Glaucoma With Blood Stasis Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015YWNL001
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Primary Open Angle Glaucoma; Drug Effect
Keywords: Primary Open Angle Glaucoma; Ginkgo biloba capsule
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test team (Active Comparator): Patients were treated with ginkgo biloba capsule regularly. Take 2 capsules 3 times a day, orally
  Interventions: Drug: Ginkgo biloba capsule
- Control group (Placebo Comparator): Patients were treated with placebo regularly.Take 2 capsules 3 times a day, orally
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ginkgo biloba capsule — Ginkgo biloba capsule may improve visual function of primary open-angle glaucoma by repairing of the optic nerve.
  Arms: Test team
Drug: Placebos — Placebos were controls.
  Arms: Control group

SUMMARY:
Primary Open Angle Glaucoma (POAG) is an eye disease that causes optic nerve damage, visual field defect, and blindness caused by increased intraocular pressure. In recent years, many studies have shown that ginkgo biloba extract has a protective effect on the visual function of glaucoma patients. Studies have shown that Ginkgo biloba capsules can improve the visual field damage of glaucoma controlled by intraocular pressure;Ginkgo biloba capsule can promote the recovery of visual evoked potential of glaucoma controlled by intraocular pressure; the improvement of visual field has a certain correlation with visual electrophysiological recovery. The mechanism may be achieved by suppressing the influx of calcium ions and thereby inhibiting the apoptosis of cells. Therefore, in this clinical study, effect of Ginkgo biloba capsule on visual function of primary open-angle glaucoma with blood stasis syndrome was evaluated by placebo as control.

DETAILED DESCRIPTION:
In this clinical study, the visual field, including MD, MS, LV, and vision score, are the main efficacy indicators. HRT and visual electrophysiological examination are the secondary efficacy indicators. Safety indicators based on laboratory tests and total frequency and incidence of adverse events. To evaluate the effectiveness and safety of Ginkgo biloba capsules for glaucoma patients with intraocular pressure control.

ELIGIBILITY:
Inclusion Criteria:

* 1. Accord with the diagnostic criteria of primary open-angle glaucoma.
* 2. Accord with the standard of blood stasis and collateralization syndrome in traditional Chinese medicine (TCM).
* 3. Intraocular pressure ≤ 18mmHg
* 4. AGIS score of visual field defect ≥ 6 points and ≤ 17 points, cup to disc ratio > 0.6, central corrected visual acuity ≥ 0.3.

Exclusion Criteria:

* 1. The diagnoses of angle closure glaucoma, absolute glaucoma, glaucoma ciliary body syndrome, high intraocular pressure (IOP) and secondary glaucoma.
* 2. Patients with various fundus diseases, such as retinal detachment, retinal vein occlusion, retinal pigmented degeneration, blood or vascular diseases.
* 3. Complicated with cornea, iris, visible lens lesion, or one-eye patient.
* 4. Patients who need to use improved circulation, nutritional nerve drugs during the trial.
* 5. Any eye surgery or laser therapy during the induction period.
* 6. Patients with a history of eye infection during the introduction period.
* 7. Complicated with severe liver and kidney diseases, or abnormal examination of liver and kidney function (ALT,AST ≥ normal upper limit 1.5 times, SCr > normal upper limit).
* 8. Complicated with severe heart and lung diseases (such as bronchial asthma or history of bronchial asthma, chronic obstructive pulmonary disease, bronchospasm, respiratory failure, etc.), diabetes, advanced tumors, blood and hematopoietic system diseases, or other serious or progressive diseases of the system.
* 9. A person who is prone to bleeding, or who has suffered severe bleeding during the period of introduction.
* 10. Pregnant, lactating women or recent birth plans.
* 11. Other conditions considered inappropriate by the investigator.
* 12. Patients who participated in other clinical trials during the introduction period.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2015-04-28 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean defect of visual field (MD) | After 48 weeks of treatment
  Detection by humphrey visual field meter

SECONDARY OUTCOMES:
Retinal nerve fiber layer thickness (RNFL) | After 12, 24, 36, and 48 weeks of treatment
  Detection by optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Ge, M.D,Ph.D, Study Chair — Zhognshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The archived documents and materials are not loaned. If the management department needs to access the original data, it should be agreed by the PI of the project.